CLINICAL TRIAL: NCT05185024
Title: A Study of Efficacy and Safety of Three Different Oral Iron-Containing Dietary Supplements in Correction of Hematological Indices and Replenishment of Depleted Iron Stores in Iron Deficient Adults With or Without Mild Microcytic Anemia
Brief Title: Daily Oral Iron Supplementation for Replenishment of Depleted Iron in Adults
Acronym: IRON-RELOAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaLinea Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: PhL-2021-IRON-RELOAD
Record Dates: First submitted 2021-12-20; First posted 2022-01-11 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Iron-deficiency; Iron Deficiency Anemia
Keywords: iron deficiency; iron supplementation; dietary supplement; >Your< Iron
MeSH Terms: conditions — Anemia, Iron-Deficiency; Iron Deficiencies | interventions — ferrous sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ferrous Sulfate Capsules (Experimental): 30 mg of elemental iron and 60 mg of vitamin C per capsule.
  Interventions: Dietary Supplement: Ferrous Sulfate Capsules; Other: Blank Liquid
- >Your< Iron Forte Capsules (Experimental): 30 mg of elemental iron and 60 mg of vitamin C per capsule.
  Interventions: Dietary Supplement: >Your< Iron Forte Capsules; Other: Blank Liquid
- >Your< Iron Forte Liquid (Experimental): 35 mg of elemental iron, 0.7 mg vitamin B6 and 1.25 mcg vitamin B12 per one dosing (5 ml).
  Interventions: Dietary Supplement: >Your< Iron Forte Liquid; Other: Blank Capsules

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate Capsules — Once daily dose of one Ferrous Sulfate Capsule for 12 weeks in total.
  Arms: Ferrous Sulfate Capsules
Dietary Supplement: >Your< Iron Forte Capsules — Once daily dose of one >Your< Iron Forte Capsule for 12 weeks in total.
  Arms: >Your< Iron Forte Capsules
Dietary Supplement: >Your< Iron Forte Liquid — Once daily dose of 5 ml of >Your< Iron Forte Liquid for 12 weeks in total.
  Arms: >Your< Iron Forte Liquid
Other: Blank Capsules — Once daily dose of one Blank Capsule (excipients only) for 12 weeks in total.
  Arms: >Your< Iron Forte Liquid
Other: Blank Liquid — Once daily dose of 5 ml of Blank Liquid (excipients only) for 12 weeks in total.
  Arms: >Your< Iron Forte Capsules; Ferrous Sulfate Capsules

SUMMARY:
The study is designed as a parallel, randomized, double blind, three-arm single-center study exploring the efficacy and safety of 12-week once daily oral dosing of iron for correction of overall iron status in 150 otherwise healthy iron-deficient adults presenting with or without mild microcytic anemia. Three iron-containing preparations in the form of either Ferrous Sulfate Capsules, >Your< Iron Forte Capsules, or >Your< Iron Forte Liquid will be tested. Potential study participants will be recruited from the general population of 18-50 year old adults. Participant eligibility will be determined by screening for hemoglobin and ferritin (in combination with C-reactive protein) levels in a sample of venous blood. Eligible individuals will be invited to participate in the study. Enrolled participants will be randomized into one of three intervention groups in a 1:1:1 ratio, receiving either Ferrous Sulfate Capsules, >Your< Iron Forte Capsules, or >Your< Iron Forte Liquid. Efficacy and safety of the assigned interventions will be evaluated through analyses of relevant hematological (hemoglobin, red blood cell indices) and biochemical (ferritin, transferrin saturation) iron-related parameters and reported adverse events after the first 4 and after a total of 12 weeks of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Personally signed and dated Informed Consent Form.
* Male or female, aged 18-50 years (inclusive) at the time of signing the Informed Consent Form.
* Iron deficiency as defined by a hemoglobin value 100-130 g/L (females) and 110-140 g/L (males) and a serum ferritin level <30 µg/L (with C-reactive protein level <10 mg/L).
* Generally healthy individual with no known significant health problems as judged by the Investigator (based on the screening questionnaire responses, medical history, the results of clinical laboratory tests performed at screening, and the results of examination of vital signs).
* Body mass index ≤27 kg/m2.
* Ability to understand and willingness to comply with all protocol required visits, assessments, and interventions.

Exclusion Criteria:

* Occult gastrointestinal bleeding (as determined by the fecal occult blood test).
* Pronounced symptoms accompanying anemia (i. e., pronounced fatigue, dizziness, shortness of breath).
* Hemochromatosis or other iron-loading disorders.
* Known hemoglobinopathy (e. g., thalassemia).
* Any active or unstable concurrent medical condition (e. g., cancer, renal dysfunction, liver dysfunction).
* Presence of an inflammatory and/or autoimmune disorder (e. g., inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, celiac disease).
* Partial or total gastrectomy or any other surgical procedure bypassing the duodenum.
* Known HIV, HBV, or HCV infection.
* Any active chronic or acute infectious disease requiring antibiotic treatment.
* Taking regular medication that could affect iron absorption (e. g., antacids, proton pump inhibitors, histamine H2 blockers).
* Use of any iron-containing medications or supplements within 30 days prior to screening and at any time throughout the duration of the study.
* Received blood transfusion within 12 weeks prior to screening or planned blood transfusion during the study period.
* Receipt of i. m. or i. v. injection of depot iron preparation within 30 days prior to screening or at any time during the study.
* Receipt of erythropoiesis stimulating agents within 30 days prior to screening or at any time during the study.
* Blood donation within the previous 30 days or planned blood donation during the study period.
* Scheduled or expected hospitalization and/or surgery during the course of the study.
* Intake of concurrent medications that could interfere with physical or mental performance (e. g., antihistamines etc.).
* For women of childbearing potential: planning of pregnancy, current pregnancy, or lactation.
* Known allergies or severe adverse reactions to previous oral iron therapy or known hypersensitivity to any component of investigational products.
* Current participation in any other interventional clinical study or participation within 30 days prior to screening.
* Any other unspecified reason (laboratory abnormality, medical condition, or psychiatric or psychological disorder) which, in the opinion of the Investigator, makes the subject unsuitable for participation in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in hemoglobin level from baseline to week 12. | 12 weeks
  Measurement in a venous blood sample.

SECONDARY OUTCOMES:
Change in hemoglobin from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in hematocrit from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in hematocrit from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular volume from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular volume from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular hemoglobin from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular hemoglobin from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular hemoglobin concentration from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in mean corpuscular hemoglobin concentration from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Change in serum ferritin level from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in serum ferritin level from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Change in transferrin saturation from baseline at week 4. | 4 weeks
  Measurement in a venous blood sample.
Change in transferrin saturation from baseline at week 12. | 12 weeks
  Measurement in a venous blood sample.
Collection and assessment of adverse events. | 4 weeks
  Collection and assessment of adverse events.
Collection and assessment of adverse events. | 12 weeks
  Collection and assessment of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Andrej Kravos, MD, PhD, Principal Investigator — Private Family Medicine Practice Andrej Kravos, MD, PhD
Locations (1):
- Diagnostic Laboratory Medicare Plus, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No